CLINICAL TRIAL: NCT03520023
Title: Does Early vs Usual Palliative Care Consultation Augment the Critical Care Physician to Decrease Healthcare Utilization and Increase Caregiver Satisfaction
Brief Title: Critical Care and Palliative Care Medicine Together in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John E. Moss, Consultant Physician, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-001107
Record Dates: First submitted 2018-04-23; First posted 2018-05-09 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Palliative Care; Intensive Care Unit; Hospice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Standard care with consultant discretion regarding consult of palliative care medicine
- Experimental (Experimental): Early palliative care consult based upon meeting study inclusion criteria
  Interventions: Other: Palliative Care Consult

INTERVENTIONS:
Other: Palliative Care Consult — Consult of hospital palliative care service for those meeting study inclusion criteria
  Arms: Experimental

SUMMARY:
Will earlier palliative care medicine consultation in the ICU result in decreased length of stay in the ICU and hospital, as well as, increased patient and family satisfaction. Secondary questions to be answered is if this early consultation changes ICU and hospital death, discharge destinations, hospice admissions, code status changes, and withdrawal of life sustaining interventions.

ELIGIBILITY:
1. Age >80 years
2. Apache II score >14
3. SOFA score > 9
4. Pre-existing functional dependency (admitted from ALF, SNF, LTAC, etc.)
5. Late stage dementia (bed-bound, nonverbal, incontinent, or unable to self-nourish/tube feed)
6. Stage 4 metastatic disease
7. Consideration to place permanent feeding tube or trach
8. Recurrent ICU admissions in the past year
9. Post-cardiac arrest
10. End-stage disease (lung, ESRD, ESLD)
11. ICU perceived need

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 1 year
  Measure will assessed by using the family satisfaction with care in the intensive care unit form (FS-ICU 24)

SECONDARY OUTCOMES:
ICU length of stay | 1 year
Ventilator Days | 1 year
Percentage admission to hospice | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John E Moss, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials